CLINICAL TRIAL: NCT03944889
Title: Quantitative Response of Healthy Muscle Following the Induction of Capsaicin
Brief Title: Quantitative Ultrasound Response of Capsaicin
Acronym: QUROC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Dinesh Kumbhare, Affiliate Scientist, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: CapsaicinUltrasound
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Central Sensitisation
Keywords: MUAP- Motor Unit Action Potential; RMS- Root Mean Square; US-Ultrasound
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Intervention Model Description: A single-centered, factorial, randomized, placebo-controlled trial with two independent variables (dosage and depth of application).
Who Masked: Participant
Masking Description: Participants and investigators will be blinded to the delivered dose; however, the type of capsaicin delivery cannot be blinded from either participants or investigators. The member of the research team conducting the randomization schedule and concealing allocation will have knowledge of and keep track of the doses contained in the containers and vials of the topical and injectable capsaicin, respectively. They will deliver the appropriate dose to the team member implementing the experimental protocol to ensure there is blinding with respect to dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (9):
- Placebo Topical (Placebo Comparator): Placebo Cream, applied topically to trapezius muscle
  Interventions: Device: Delsys Trigno Galileo System; Device: Cadwell Sierra Wave; Device: Sonosite Ultrasound Machine; Device: Goniometer
- Low Dose, Topical (Active Comparator): Capsaicin Cream- low dosage, applied topically to trapezius
  Interventions: Drug: Capsaicin; Device: Delsys Trigno Galileo System; Device: Cadwell Sierra Wave; Device: Sonosite Ultrasound Machine; Device: Goniometer
- High Dose, Topical (Active Comparator): Capsaicin Cream- higher dosage, applied topically to trapezius
  Interventions: Drug: Capsaicin; Device: Delsys Trigno Galileo System; Device: Cadwell Sierra Wave; Device: Sonosite Ultrasound Machine; Device: Goniometer
- Placebo, Intrafascial (Placebo Comparator): Injection placebo(saline)- injected intrafascially into trapezius
  Interventions: Device: Delsys Trigno Galileo System; Device: Cadwell Sierra Wave; Device: Sonosite Ultrasound Machine; Device: Goniometer
- Low Dose, Intrafacial (Active Comparator): Injection Capsaicin formulation low dose- injected intrafascially into trapezius
  Interventions: Drug: Capsaicin; Device: Delsys Trigno Galileo System; Device: Cadwell Sierra Wave; Device: Sonosite Ultrasound Machine; Device: Goniometer
- High Dose, Intrafascial (Active Comparator): Injection Capsaicin formulation higher dose- injected intrafascially into trapezius
  Interventions: Drug: Capsaicin; Device: Delsys Trigno Galileo System; Device: Cadwell Sierra Wave; Device: Sonosite Ultrasound Machine; Device: Goniometer
- Placebo, Intramuscular (Placebo Comparator): Injection placebo (saline) - injected intramuscularly into trapezius
  Interventions: Device: Delsys Trigno Galileo System; Device: Cadwell Sierra Wave; Device: Sonosite Ultrasound Machine; Device: Goniometer
- Low Dose, Intramuscular (Active Comparator): Injection Capsaicin formulation low dose - injected intramuscularly into trapezius
  Interventions: Drug: Capsaicin; Device: Delsys Trigno Galileo System; Device: Cadwell Sierra Wave; Device: Sonosite Ultrasound Machine; Device: Goniometer
- High Dose, Intramuscular (Active Comparator): Injection Capsaicin formulation higher dose - injected intramuscularly into trapezius
  Interventions: Drug: Capsaicin; Device: Delsys Trigno Galileo System; Device: Cadwell Sierra Wave; Device: Sonosite Ultrasound Machine; Device: Goniometer

INTERVENTIONS:
Drug: Capsaicin — Capsaicin 50ug (low dose), Capsaicin 100ug(high dose) will be administered as a topical skin cream and will be intermixed with saline for the injectable solution.
  Arms: High Dose, Intrafascial; High Dose, Intramuscular; High Dose, Topical; Low Dose, Intrafacial; Low Dose, Intramuscular; Low Dose, Topical
Device: Delsys Trigno Galileo System — This device is a wireless surface EMG device.
Device: Cadwell Sierra Wave — Intramuscular EMG recording machinery
Device: Sonosite Ultrasound Machine — Ultrasound System
Device: Goniometer — A device to measure angular position

SUMMARY:
Central Sensitization is an aspect of chronic pain and is associated with over-excitability of the central nervous system. Central Sensitization normally presents itself with other chronic syndromes such as Myofascial Pain Syndrome, so it is difficult to separate the characteristics of the two. The purpose of this study is to determine whether sensitizing healthy muscle using capsaicin, a chilli pepper extract, induces a regional change in ultrasound texture features of the targeted muscle, or the muscles in that are in close proximity. This regional change will be accompanied by electromyography (EMG) recordings to confirm the presence of abnormality. Topical capsaicin and injectable capsaicin will be applied at three different concentrations, 0ug(placebo effect),50ug and 100ug.

Research Questions:

Does sensitization cause a significant regional change in the texture features of the targeted muscle or surrounding muscles? Is this regional change confirmed by abnormality of motor unit firing rates or EMG amplitudes? Is the response dose dependent? Does the induced central sensitization cause a change in force steadiness?

Experimental Protocol:

The physician on site will apply surface and intramuscular EMG sensors to the trapezius. A goniometer will be placed on the subjects arm to detect position. Following this, an ultrasound image of the trapezius, supraspinatus and infraspinatus will be taken.The participant will perform an increasing and decreasing contraction.The subject will then have capsaicin injected into their trapezius or applied onto their skin. The exercise and measurements will then be repeated. The ultrasound will be acquired by the Sonosite ultrasound system. The EMG data will be acquired by the Delsys Trigno EMG system for the surface EMG and the Cadwell Sierra Wave system for the intramuscular EMG. The data will be processed through Delsys EMGworks software and MATLAB. Texture features of the pre and post injection ultrasound images will be compared. Decomposition of motor units will allow for the analysis of motor unit action potential firing rate and amplitudes. Analysis of force steadiness will also be calculated via the goniometer.

Overall, the findings from this study should present preliminary evidence to inform central sensitization's effects on regional muscle structure changes, functional changes and motor unit activity.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is a prevalent chronic pain disorder primarily characterized by myofascial trigger points (MTrP). There is limited knowledge on the pathophysiology and mechanisms underlying MTrP and its development. Ultrasound investigations that have been performed on trigger points can differentiate between active and latent trigger points, but have not characterized the central sensitization aspect of them. The electromyography (EMG) investigations of central sensitization that have been performed mostly use hypertonic saline to induce hyperalgesia, and have demonstrated conflicting results. Central sensitization has been proposed as the primary mechanism underlying MTrP development. Central sensitization is associated with hyperexcitability of neuronal responses to normal or noxious stimuli. There is a need for a study that quantifies regional central sensitization using ultrasound to measure the changing structure, and electromyography to measure specific motor unit activity responses in the muscle.

Purpose The purpose of this study is to determine whether sensitizing healthy muscle using capsaicin induces a change in the structural integrity of the affected muscle, and determine if the motor unit frequency and amplitudes change within that region. Central sensitization will be induced using topical capsaicin and injectable capsaicin at three different concentrations. This is an exploratory trial that aims to provide preliminary evidence on whether central sensitization is a direct cause of taut band and MTrP development.

Our specific research questions are followings:

1. Does sensitization cause a significant regional change in the texture features of the targeted muscle or surrounding muscles?
2. Does capsaicin induced sensitization elicit a change in motor unit action potential(MUAP) amplitude by approximately 20 to 25% within the region of experimentally induced central sensitization or in the region of texture feature changes? Our hypothesis for this portion of the study is that sensitization modifies the anterior horn cell activity which will be measured by the amplitude of the potentials.
3. Does capsaicin induced sensitization elicit continuous electrical activity as observed in MTrPs? This tests the hypothesis that sensitization creates the presence of continuous low amplitude action potentials.
4. Does capsaicin induced sensitization influence the rate of recruitment of motor units in the muscle within the region induced? Does this occur within the regions identified by the changes in texture features? The recruitment of motor units is normally expected to follow the Henneman size principle.[20-23] Our hypothesis for this portion of the study is that sensitization will cause an aberration in recruitment. If this is demonstrated, then there is modification of the normal processing at both dorsal and ventral horns of the spinal cord.
5. Is there a location dependent EMG response to capsaicin induced sensitization? In other words, do the texture features or EMG responses from muscles that lie anatomically distant from the location of the site of intramuscular capsaicin injection have changes from their baseline calculations? This would test the hypothesis that type III and IV afferents have an influence on the anterior horn cells that lie distant to the ones that are supplying muscle fibers in the vicinity of the stimulated sensory afferents.
6. Is there a dose dependent EMG response at motor units to capsaicin induced sensitization? Here, the hypothesis of causality will be assessed in a preliminary manner. If there is a relationship then further experiments that more thoroughly assess causality will be needed.

This proposed study is a single centered, factorial, randomized placebo-controlled trial with two independent variables, depth of capsaicin application(3 levels) and dose of capsaicin(3 levels), for a total of 6 treatment arms and three control groups.The first between groups variable will be topical capsaicin application, injectable(intrafascial) and injectable(intramuscular) capsaicin injection. Within each partition, there will be three treatments: control, 50 micrograms, 100 micrograms. The control group will receive a topical skin lotion that is inert and has no sensitization effect. An equal number of participants will be allocated to each of the six treatment groups using an electronic randomization generator. Block randomization will be used to ensure equal allotment into each group.

Capsaicin Application and Injection Capsaicin will be applied directly to the region of the innervation zone at the muscle belly to sensitize the neurons within the region of taut band development. Topical and intramuscular capsaicin will be used. The capsaicin formula will be compounded by a registered pharmacist. Topical capsaicin will be delivered in a cream and injectable capsaicin will be intermixed with saline prior to injection. The control group in the topical capsaicin arm will be treated with the cream base used during the experiment without added capsaicin and the injection arm will be injected with saline. A trained medical professional on the research team will apply the topical capsaicin or topical placebo treatments. The region of topical application will measure 5cm squared in the dermatome zone location to cover an area of approximately 25cm2. A trained physician in physical medicine and rehabilitation will deliver injectable capsaicin using a 27-gauge needle at the location of the superior fascia of the upper trapezius muscle with ultrasound guidance. Intramuscular capsaicin will also be injected using ultrasound guidance to avoid the superior or inferior fascia.

To confirm the presence of central sensitization, brush allodynia will be used to detect mechanical hyperalgesia outside the region of primary nociception. The size of the region of secondary hyperalgesia will be measured to characterize the extent of central sensitization. This will be accomplished using a tape measure and the perpendicular dimensions of the region of secondary hyperalgesia will be recorded in square centimeters.

Experimental Protocol The anatomical location for ultrasound probe and electrode placement will be identified for each participant. The ultrasound probe will be placed on 3 muscles: the trapezius, the supraspinatus, and the infraspinatus. Two ultrasonic pictures will be taken of each. The area will then be cleaned with alcohol and water. The Delsys Galileo sensor, and the intramuscular needle electrode will be placed directly on the trapezius' identified area. Participants will be asked to gently contract their trapezius muscle. They will be instructed to perform a gradually increasing contraction in isometric condition, in a controlled manner. They will hold this contraction at 30% of their maximal voluntary contraction, and then perform a gradually decreasing contraction to rest. This will be performed four times for each type of study intervention and before as well as after each intervention, namely topical control cream, topical capsaicin at 50ug and 100 ug, injection of the superior aspect of the superior fascia followed by intramuscular injection with these two concentrations of capsaicin. The placement of these latter will be verified by ultrasound guidance. The intramuscular needle will then be removed and participants will be bandaged and cared for appropriately by the expert physician performing the experiment. Participants will be re-examined to determine if there were any adverse effects from the experimental procedures. If any occurred, then these will be carefully managed by the medical members of the research team and recorded. Participants will be asked to remain at the lab for an additional 30 minutes to ensure they are well prior to leaving.

Ultrasound Analysis Texture analysis will be performed using MATLAB and the image and signal processing toolbox. Analyses will include first order parameters such as mean and standard deviation of the pixel level values, as well as second order parameters, which provide details on the spatial distribution of pixel values. These include co-occurance and run-length matrices, local binary pattern and blob analysis.

EMG Analysis The following parameters will be analyzed: the firing times and frequency of individual motor units, motor unit action potential amplitude and shapes, the root mean square value (RMS) of each channel and of the entire signal, the coefficient of variation for force steadiness, and the centroid of the EMG signal in the cranial-caudal and the medial-lateral directions. These procedures will be repeated for each contraction.

The results of this study should provide insight into the structural changes and motor changes at the region of sensitization, as well as in adjacent muscles.This will provide further insight as to whether structural changes are accompanied by motor changes within the same region, and inform further investigations into the pathophysiology of myofascial pain.

The full study protocol and statistical analysis plan is submitted in the documents section.

ELIGIBILITY:
Inclusion Criteria:

* healthy with no past medical history
* a visual analogue score below 3 indicating low pain severity, ideally who complain of no pain
* right or left handed
* normal body mass index
* have sufficient knowledge of the English language to provide informed consent and understand the protocols
* agree to sign a consent form.

Exclusion Criteria:

* history of pain
* detectable myofascial trigger points upon physical examination
* history of pain related disturbances such as poor sleep
* cognitive disturbances, psychiatric disorders
* history of general medical disorder that may affect the outcome of the study such as diabetes mellitus
* history of cervical radiculopathies
* history of inflammatory arthropathy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Motor Unit Action Potential Firing Rate | up to 6 months
  Firing rate will be determined using EMGworks software and compared with baseline firing rates.
Root Mean Square EMG values | up to 6 months
  Root mean square values will be compared with baseline values using EMGworks software.
Coefficient of Variation- Force steadiness | up to 6 months
  Force steadiness will be measured by the coefficient of variation (standard deviation/mean) using EMGworks software, validated through the goniometer measurements
Motor Unit Action Potential Amplitudes | up to 6 months
  Amplitudes will be measured from the overall amplitude difference from baseline for each motor unit using EMGworks software
Centroid of Frequency Spectrum | up to 6 months
  Centroid frequency will be measured and the frequency shift of the signal will be compared with baseline. Measured using EMGworks software
Texture Feature Analysis | up to 6 months
  91 features will be extracted using MATLAB, then a reduction of variables will be performed using principal component analysis. The experimental data will be compared with baseline results.

SECONDARY OUTCOMES:
Severity of pain | up to 6 months
  Pain, or burning sensation measured by the visual analogue scale(0-no pain to 10-worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh M Kumbahre, MD,PhD, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The University Health Network has a high importance on patient confidentiality. For ethics approval, this was complied with these standards, upholding the patient confidentiality standard at UHN.

REFERENCES:
- [Background] Srbely JZ. New trends in the treatment and management of myofascial pain syndrome. Curr Pain Headache Rep. 2010 Oct;14(5):346-52. doi: 10.1007/s11916-010-0128-4. PMID 20607458
- [Background] Masuda T, Sadoyama T. Distribution of innervation zones in the human biceps brachii. J Electromyogr Kinesiol. 1991 Jun;1(2):107-15. doi: 10.1016/1050-6411(91)90004-O. PMID 20870500
- [Background] Barbero M, Cescon C, Tettamanti A, Leggero V, Macmillan F, Coutts F, Gatti R. Myofascial trigger points and innervation zone locations in upper trapezius muscles. BMC Musculoskelet Disord. 2013 Jun 8;14:179. doi: 10.1186/1471-2474-14-179. PMID 23758854
- [Background] Melzack R, Stillwell DM, Fox EJ. Trigger points and acupuncture points for pain: correlations and implications. Pain. 1977 Feb;3(1):3-23. doi: 10.1016/0304-3959(77)90032-X. PMID 69288
- [Background] Hong CZ, Simons DG. Pathophysiologic and electrophysiologic mechanisms of myofascial trigger points. Arch Phys Med Rehabil. 1998 Jul;79(7):863-72. doi: 10.1016/s0003-9993(98)90371-9. PMID 9685106
- [Background] Gerwin RD, Dommerholt J, Shah JP. An expansion of Simons' integrated hypothesis of trigger point formation. Curr Pain Headache Rep. 2004 Dec;8(6):468-75. doi: 10.1007/s11916-004-0069-x. PMID 15509461
- [Background] Bron C, Dommerholt JD. Etiology of myofascial trigger points. Curr Pain Headache Rep. 2012 Oct;16(5):439-44. doi: 10.1007/s11916-012-0289-4. PMID 22836591
- [Background] Yu SH, Kim HJ. Electrophysiological characteristics according to activity level of myofascial trigger points. J Phys Ther Sci. 2015 Sep;27(9):2841-3. doi: 10.1589/jpts.27.2841. Epub 2015 Sep 30. PMID 26504306
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Graven-Nielsen T, Arendt-Nielsen L. Assessment of mechanisms in localized and widespread musculoskeletal pain. Nat Rev Rheumatol. 2010 Oct;6(10):599-606. doi: 10.1038/nrrheum.2010.107. Epub 2010 Jul 27. PMID 20664523
- [Background] Fernandez-de-las-Penas C, Cuadrado ML, Arendt-Nielsen L, Simons DG, Pareja JA. Myofascial trigger points and sensitization: an updated pain model for tension-type headache. Cephalalgia. 2007 May;27(5):383-93. doi: 10.1111/j.1468-2982.2007.01295.x. Epub 2007 Mar 14. PMID 17359516
- [Background] Kim Y, Kim J, Shim JK, Suh DW, Yoon B. The hypoalgesic effect of remote tactile sensory modulation on the mechanical sensitivity of trigger points: A randomized controlled study. NeuroRehabilitation. 2014;35(3):607-14. doi: 10.3233/NRE-141156. PMID 25248449
- [Background] LaMotte RH, Lundberg LE, Torebjork HE. Pain, hyperalgesia and activity in nociceptive C units in humans after intradermal injection of capsaicin. J Physiol. 1992 Mar;448:749-64. doi: 10.1113/jphysiol.1992.sp019068. PMID 1593488
- [Background] Srbely JZ, Dickey JP, Bent LR, Lee D, Lowerison M. Capsaicin-induced central sensitization evokes segmental increases in trigger point sensitivity in humans. J Pain. 2010 Jul;11(7):636-43. doi: 10.1016/j.jpain.2009.10.005. Epub 2009 Dec 16. PMID 20015704
- [Background] Torebjork HE, Lundberg LE, LaMotte RH. Central changes in processing of mechanoreceptive input in capsaicin-induced secondary hyperalgesia in humans. J Physiol. 1992 Mar;448:765-80. doi: 10.1113/jphysiol.1992.sp019069. PMID 1593489
- [Background] Dideriksen JL, Holobar A, Falla D. Preferential distribution of nociceptive input to motoneurons with muscle units in the cranial portion of the upper trapezius muscle. J Neurophysiol. 2016 Aug 1;116(2):611-8. doi: 10.1152/jn.01117.2015. Epub 2016 May 25. PMID 27226455
- [Background] Falla D, Farina D. Motor units in cranial and caudal regions of the upper trapezius muscle have different discharge rates during brief static contractions. Acta Physiol (Oxf). 2008 Apr;192(4):551-8. doi: 10.1111/j.1748-1716.2007.01776.x. Epub 2007 Nov 2. PMID 17979997
- [Background] Lee U, Kim M, Lee K, Kaplan CM, Clauw DJ, Kim S, Mashour GA, Harris RE. Functional Brain Network Mechanism of Hypersensitivity in Chronic Pain. Sci Rep. 2018 Jan 10;8(1):243. doi: 10.1038/s41598-017-18657-4. PMID 29321621
- [Background] Schmidt-Wilcke T, Clauw DJ. Fibromyalgia: from pathophysiology to therapy. Nat Rev Rheumatol. 2011 Jul 19;7(9):518-27. doi: 10.1038/nrrheum.2011.98. PMID 21769128
- [Background] HENNEMAN E, SOMJEN G, CARPENTER DO. FUNCTIONAL SIGNIFICANCE OF CELL SIZE IN SPINAL MOTONEURONS. J Neurophysiol. 1965 May;28:560-80. doi: 10.1152/jn.1965.28.3.560. No abstract available. PMID 14328454
- [Background] Ertas M, Stalberg E, Falck B. Can the size principle be detected in conventional EMG recordings? Muscle Nerve. 1995 Apr;18(4):435-9. doi: 10.1002/mus.880180410. PMID 7715629
- [Background] Vilensky JA, Gilman S. Renaming the "Henneman size principle". Science. 1998 Jun 26;280(5372):2031. doi: 10.1126/science.280.5372.2027f. No abstract available. PMID 9669955
- [Background] Szolcsanyi J. A pharmacological approach to elucidation of the role of different nerve fibres and receptor endings in mediation of pain. J Physiol (Paris). 1977 Sep;73(3):251-9. PMID 926026
- [Background] Carpenter SE, Lynn B. Vascular and sensory responses of human skin to mild injury after topical treatment with capsaicin. Br J Pharmacol. 1981 Jul;73(3):755-8. doi: 10.1111/j.1476-5381.1981.tb16812.x. PMID 6166346
- [Background] Simone DA, Baumann TK, LaMotte RH. Dose-dependent pain and mechanical hyperalgesia in humans after intradermal injection of capsaicin. Pain. 1989 Jul;38(1):99-107. doi: 10.1016/0304-3959(89)90079-1. PMID 2780068
- [Background] Ishimaru K, Kawakita K, Sakita M. Analgesic effects induced by TENS and electroacupuncture with different types of stimulating electrodes on deep tissues in human subjects. Pain. 1995 Nov;63(2):181-187. doi: 10.1016/0304-3959(95)00030-V. PMID 8628583
- [Background] Langevin HM, Fox JR, Koptiuch C, Badger GJ, Greenan-Naumann AC, Bouffard NA, Konofagou EE, Lee WN, Triano JJ, Henry SM. Reduced thoracolumbar fascia shear strain in human chronic low back pain. BMC Musculoskelet Disord. 2011 Sep 19;12:203. doi: 10.1186/1471-2474-12-203. PMID 21929806
- [Background] Schilder A, Hoheisel U, Magerl W, Benrath J, Klein T, Treede RD. Sensory findings after stimulation of the thoracolumbar fascia with hypertonic saline suggest its contribution to low back pain. Pain. 2014 Feb;155(2):222-231. doi: 10.1016/j.pain.2013.09.025. Epub 2013 Sep 26. PMID 24076047
- [Background] Barbero M, Gatti R, Lo Conte L, Macmillan F, Coutts F, Merletti R. Reliability of surface EMG matrix in locating the innervation zone of upper trapezius muscle. J Electromyogr Kinesiol. 2011 Oct;21(5):827-33. doi: 10.1016/j.jelekin.2011.05.013. Epub 2011 Jul 12. PMID 21752668
- [Background] Kumbhare D, Shaw S, Grosman-Rimon L, Noseworthy MD. Quantitative Ultrasound Assessment of Myofascial Pain Syndrome Affecting the Trapezius: A Reliability Study. J Ultrasound Med. 2017 Dec;36(12):2559-2568. doi: 10.1002/jum.14308. Epub 2017 Jul 3. PMID 28670779
- [Background] Kumbhare DA, Ahmed S, Behr MG, Noseworthy MD. Quantitative Ultrasound Using Texture Analysis of Myofascial Pain Syndrome in the Trapezius. Crit Rev Biomed Eng. 2018;46(1):1-31. doi: 10.1615/CritRevBiomedEng.2017024947. PMID 29717675
- [Background] Farina D, Madeleine P, Graven-Nielsen T, Merletti R, Arendt-Nielsen L. Standardising surface electromyogram recordings for assessment of activity and fatigue in the human upper trapezius muscle. Eur J Appl Physiol. 2002 Apr;86(6):469-78. doi: 10.1007/s00421-001-0574-0. Epub 2002 Feb 19. PMID 11944093
- [Background] Holobar A, Zazula D. Correlation-based decomposition of surface electromyograms at low contraction forces. Med Biol Eng Comput. 2004 Jul;42(4):487-95. doi: 10.1007/BF02350989. PMID 15320457
- [Background] Holobar A, Zazula D. Multichannel blind source separation using convolution kernel compensation. IEEE Transactions on Signal Processing 2007;55(9):4487-96.
- [Background] Henneman E, Mendell LM. Functional organization of motoneuron pool and its inputs. Handbook of Physiology. The Nervous System. Motor Control. 1981;1:423-507
- [Background] Holobar A, Farina D, Gazzoni M, Merletti R, Zazula D. Estimating motor unit discharge patterns from high-density surface electromyogram. Clin Neurophysiol. 2009 Mar;120(3):551-62. doi: 10.1016/j.clinph.2008.10.160. Epub 2009 Feb 8. PMID 19208498
- [Background] Holobar A, Minetto MA, Botter A, Negro F, Farina D. Experimental analysis of accuracy in the identification of motor unit spike trains from high-density surface EMG. IEEE Trans Neural Syst Rehabil Eng. 2010 Jun;18(3):221-9. doi: 10.1109/TNSRE.2010.2041593. Epub 2010 Feb 8. PMID 20144921
- [Background] Holobar A, Glaser V, Gallego JA, Dideriksen JL, Farina D. Non-invasive characterization of motor unit behaviour in pathological tremor. J Neural Eng. 2012 Oct;9(5):056011. doi: 10.1088/1741-2560/9/5/056011. Epub 2012 Sep 10. PMID 22962251
- [Background] Bandholm T, Rasmussen L, Aagaard P, Diederichsen L, Jensen BR. Effects of experimental muscle pain on shoulder-abduction force steadiness and muscle activity in healthy subjects. Eur J Appl Physiol. 2008 Apr;102(6):643-50. doi: 10.1007/s00421-007-0642-1. Epub 2007 Dec 8. PMID 18066578
- [Background] Huynh H, Feldt LS. Estimation of the Box correction for degrees of freedom from sample data in randomized block and split-plot designs. J Edu Stat 1976;1(1):69-82
- [Background] Shah JP, Gilliams EA. Uncovering the biochemical milieu of myofascial trigger points using in vivo microdialysis: an application of muscle pain concepts to myofascial pain syndrome. J Bodyw Mov Ther. 2008 Oct;12(4):371-384. doi: 10.1016/j.jbmt.2008.06.006. Epub 2008 Aug 13. PMID 19083696
- [Background] Falla D, Farina D, Graven-Nielsen T. Experimental muscle pain results in reorganization of coordination among trapezius muscle subdivisions during repetitive shoulder flexion. Exp Brain Res. 2007 Apr;178(3):385-93. doi: 10.1007/s00221-006-0746-6. Epub 2006 Oct 19. PMID 17051373
- [Background] Mclean L, Urquhart N. The influence of psychological stressors on myoelectrical signal activity in the shoulder region during a data entry task. Work Stress 2002;16(2):138-53
- [Background] Westad C. Motor control of the upper trapezius. 2005
- [Derived] Evans V, Behr M, Masani K, Kumbhare D. Quantitative response of healthy muscle following the induction of capsaicin: an exploratory randomized controlled trial. Trials. 2020 Dec 11;21(1):1020. doi: 10.1186/s13063-020-04937-4. PMID 33308274

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT03944889/Prot_SAP_002.pdf